CLINICAL TRIAL: NCT05515679
Title: The BRAIN App: Building Relationships Using Artificial Intelligence and Nostalgia
Acronym: BRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopeful Aging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R43AG071105-01A1 (NIH)
Record Dates: First submitted 2022-08-10; First posted 2022-08-25 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Dementia; Dementia, Vascular; Alzheimer Disease; Dementia, Mixed
Keywords: psychosocial; non-pharmacological
MeSH Terms: conditions — Dementia; Dementia, Vascular; Alzheimer Disease; Mixed Dementias

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): BRAIN Intervention
  Interventions: Behavioral: The BRAIN App

INTERVENTIONS:
Behavioral: The BRAIN App — The BRAIN App will be the first-ever artificial intelligence enabled cognitive stimulation therapy app, specifically designed for PWD. The goal of the app is to foster positive relationships between the care triad.

SUMMARY:
This study will involve testing of an Alpha version of an app called "Building Relationships using Artificial Intelligence and Nostalgia" or BRAIN. The BRAIN App will be the first -ever artificial intelligence infused CST app for PWD. The app has two main goals: (1) to foster positive relationships between the care triad, and (2) to promote QoL while reducing responsive behaviors in PWD. Testing will examine the app's impact on engagement/affect for both PWD and professional Care Partners.

DETAILED DESCRIPTION:
A quasi-experimental pretest / posttest design will be used. During a four-week baseline period, researchers will collect data on engagement, quality of life, neuropsychiatric symptoms, and quality of the care-patient relationship. Participants will then use the BRAIN app for four weeks, during which engagement data will be collect. After the intervention period, researchers will collect data again on quality of life, neuropsychiatric symptoms, and quality of the carer-patient relationship.

ELIGIBILITY:
PWD Inclusion Criteria:

* diagnosed with dementia (any type)
* resident in ALF or NH
* 65+ years old
* read and speak English
* exhibit at least one responsive behavior on the NPI-NH or score below maximum score on the DEMQOL

PWD Exclusion Criteria:

* bed-confined
* completely unable to communicate verbally
* have serious visual or hearing impairments
* show signs of rapid decline or over the last six months

Staff and Family Member Inclusion Criteria

* 18+ years old
* speak and read English

Staff and Family Member Exclusion Criteria

-n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Skrajner, MA, Principal Investigator — Hopeful Aging
Locations (1):
- The Hearthstone Institute, Winchester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Persons With Dementia: Persons with dementia (PWD) were the "primary" or "target" participants in the study. PWD participated by initially participating in baseline interviews. Then, the person was invited to participate in the BRAIN intervention twice per week for five weeks.
- Staff Members: Staff members participated by providing feedback on the app and training. In addition, staff took pre- and post-quizzes for the training.
- Family Members: Family members exclusively participated by providing information about their loved one's (i.e., person with dementia's) background, interests and preferences. Please note: although we originally expected one family some persons with dementia did not have a family member available who could be contacted regarding their background, interests, and preferences. As such, the total number of family members is not equal to the persons with dementia. When a family member want not available, information about the person with dementia was obtained by the person with dementia himself or herself.
Period: Baseline
Arm/Group | Persons With Dementia | Staff Members | Family Members
Started | 22 | 13 | 10
Completed | 22 | 13 | 10
Not Completed | 0 | 0 | 0
Period: Treatment
Arm/Group | Persons With Dementia | Staff Members | Family Members
Started | 22 | 13 | 0 (family members had no involvement in the treatment period.)
Completed | 22 | 13 | 0 (family members were not involved in the treatment period.)
Not Completed | 0 | 0 | 0
Period: Post-Treatment
Arm/Group | Persons With Dementia | Staff Members | Family Members
Started | 22 | 13 | 0 (family members were not involved in post-treatment.)
Completed | 22 | 13 | 0 (family members were not involved in post-treatment.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Family Members: Family members exclusively participated by providing information about their loved one's (i.e., person with dementia's) background, interests and preferences. As such, there is no outcome data for family members. Please note: although we originally expected one family some persons with dementia did not have a family member available who could be contacted regarding their background, interests, and preferences. As such, the total number of family members is not equal to the persons with dementia. When a family member want not available, information about the person with dementia was obtained by the person with dementia himself or herself.
- Total: Total of all reporting groups
Arm/Group | Persons With Dementia | Staff Members | Family Members | Total
Number analyzed (Participants) | 22 | 13 | 10 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 13 | 6 | 19
  >=65 years | 22 | 0 | 4 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.73 (6.53) | 45.92 (11.67) | 65.00 (11.1) | 68.6 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 6 | 33
  Male | 8 | 0 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 12 | 10 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 0 | 9
  White | 16 | 10 | 10 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 13 | 10 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Treatment for Constructive Engagement on the Menorah Park Engagement Scale
Description: Constructive Engagement on the Menorah Park Engagement Scale is defined as doing or commenting on something related to the target activity. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple BRAIN activities were observed and a mean was calculated. The minimum value for Constructive Engagement is zero (0) and the maximum score is two (2). Higher scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | .72 (.48)
Statistical Analysis 1: Comparison: Persons With Dementia; Using a paired sample t-test (two tailed), we wished to examine whether there was an increase in Constructive Engagement and Pleasure and a reduction in Passive Engagement, Distracted Engagement, and Non-Engagement, from baseline to treatment. With an anticipated PWD sample of 24, and using means and standard deviations from the PI's previous studies, we calculated a power of 90% to detect effects (alpha = .05; one-tailed test). (3) PWD and staff report high satisfaction wi; Test type: Superiority; p < 0.01, t-test, 2 sided; Median Difference (Final Values) = 0.72, 95% CI 2-sided [.51 to .94], Standard Deviation .48

2. Primary Outcome: Change From Baseline to Treatment for Passive Engagement on the Menorah Park Engagement Scale
Description: Passive Engagement on the Menorah Park Engagement Scale is defined as listening or watching something related to the target activity. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple BRAIN activities were observed and a mean was calculated. The minimum value for Passive Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | -0.33 (.60)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p = .017, t-test, 2 sided; Mean Difference (Final Values) = -.33, 95% CI 2-sided [-0.59 to -0.07], Standard Deviation .60

3. Primary Outcome: Change From Baseline to Treatment for Other Engagement on the Menorah Park Engagement Scale
Description: Other Engagement on the Menorah Park Engagement Scale is defined as doing, commenting, listening, or watching something NOT related to the target activity. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple BRAIN activities were observed and a mean was calculated. The minimum value for Other Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | -.25 (.40)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p = .008, t-test, 2 sided; Mean Difference (Final Values) = -.25, 95% CI 2-sided [-0.43 to -0.07], Standard Deviation .41

4. Primary Outcome: Change From Baseline to Treatment for Non-Engagement on the Menorah Park Engagement Scale
Description: Non-Engagement on the Menorah Park Engagement Scale is defined as sleeping and/or staring into space. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple BRAIN activities were observed and a mean was calculated. The minimum value for Non-Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | -0.15 (.34)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p = 0.053, t-test, 2 sided; Median Difference (Final Values) = -.15, 95% CI 2-sided [-.30 to -.00], Standard Deviation 0.34

5. Primary Outcome: Change From Baseline to Treatment for Pleasure on the Menorah Park Engagement Scale
Description: Pleasure on the Menorah Park Engagement Scale is defined as clearly observable laughing or smiling. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple BRAIN activities were observed and a mean was calculated. The minimum value for Pleasure is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | .66 (.28)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p < .01, t-test, 2 sided; Mean Difference (Final Values) = .66, 95% CI 2-sided [.54 to .79], Standard Deviation .28

6. Primary Outcome: Change From Baseline to Treatment for Positive Items Sub-score on the Engagement of Persons With Dementia Scale (EPWDS)
Description: The Positive Items Sub-score on the EPWDS is the total score for the five following items: (1) Displays positive affect, (2) maintains eye contact, (3) Initiates, participates, or maintains verbal conversation, sounds or gestures (e.g., nodding) in response to the activity, or the materials used, or the person/s involved, (4) Responds to an activity by approaching, reaching out, touching, holding or handling the activity, the material used, or the person/s involved, and (5) Uses the activity or the material/s to encourage others to interact, or as a communication channel to interact and talk with others (e.g., staff and other residents). During baseline, multiple observations of "standard" activities were observed and a mean was calculated for the positive item sub-score. Then, again, during treatment, multiple BRAIN activities were observed and a mean was calculated. The minimum value is 0 and the maximum score is 20. Higher scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | 4.11 (3.35)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 4.11, 95% CI 2-sided [2.62 to 5.60], Standard Deviation 3.35

7. Primary Outcome: Change From Baseline to Treatment for Negative Items Sub-score on the Engagement of Persons With Dementia Scale (EPWDS)
Description: The Negative Items Sub-score on the EPWDS is the total score for the five following items: (1) Displays negative affect, (2) Appears inattentive, has an unfocused stare or turns head/eyes away from the activity, materials used, or the person/s involved, (3) Refuses to participate in the activity or in a conversation related to the activity by verbalizing e.g. "no", "stop", etc. OR verbalizes negative comment, complaint, and sound in response to or related to the activity, or the materials used, or the person/s involved, and (4) In response to the activity, is distracting or disrupting others (e.g., Staff/facilitator and other residents). During baseline, multiple observations of "standard" activities were observed and a mean was calculated for the negative item sub-score. Then, again, during treatment, multiple observations were taken and mean was calculate. Total score ranges from 0 to 16. Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | -1.07 (1.10)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-1.55 to -0.58], Standard Deviation 1.10

8. Secondary Outcome: Change From Baseline to Treatment on Dementia Related Quality of Life (DEMQOL)
Description: The Dementia Related Quality of Life Scale is a 28 item scale that examines quality of life in persons with dementia. The score ranges for 28 to 112. Higher scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | 6.02 (11.4)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p = .022, t-test, 2 sided; Median Difference (Final Values) = 6.02, 95% CI 2-sided [0.97 to 11.1], Standard Deviation 11.4

9. Secondary Outcome: Change From Baseline to Treatment on the Neuropsychiatric Inventory-Nursing Home (NPI-NH), Frequency x Severity Score (FxS)
Description: The NPI-NH examines 10 types of neuropsychiatric symptoms in persons with dementia, with the FxS score looking creating a composite score that takes into account frequency and severity of the symtoms. The score ranges from 0 to 120. Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia
Number analyzed (Participants) | 22
score on scale | 1.23 (9.5)
Statistical Analysis 1: Comparison: Persons With Dementia; Test type: Superiority; p = .551, t-test, 2 sided; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-2.90 to 5.44], Standard Deviation 9.50

10. Secondary Outcome: Change From Pre-Test to Post-Test for the Knowledge Assessment for BRAIN Training for Staff
Description: Staff took a quiz at pre-test and again at post-test. Scores range from 0 to 100, with higher scores representing a better outcome
Time Frame: Baseline (Week 1) and Post-Training (Week 5)
Measure: Mean (Standard Deviation); unit: percent score on quiz out of 100
Groups:
- Staff Members: Staff members participated by providing feedback on the app and training. In addition, staff took pre and post quizzes for the BRAIN Training.
Arm/Group | Staff Members
Number analyzed (Participants) | 13
percent score on quiz out of 100 | 27.43 (.11)
Statistical Analysis 1: Comparison: Staff Members; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 27.43, 95% CI 2-sided [17.7 to 37.2], Standard Deviation 0.11

11. Secondary Outcome: Percent of Staff Who Thought Residents Enjoyed BRAIN Activities
Description: Staff were asked if they thought residents enjoyed using the BRAIN Activities. The total who said YES was converted into a percentage. Total score ranges from 0 to 100, with higher scores representing a better outcome.
Time Frame: Post-Treatment (Week 11)
Measure: Number; unit: percentage who said yes
Arm/Group | Staff Members
Number analyzed (Participants) | 12
percentage who said yes | 100

12. Secondary Outcome: Percent of Staff Who Said They Would Recommend the BRAIN App to Colleagues
Description: Staff were asked if they would recommend BRAIN Activities to colleagues. The total who said YES was converted into a percentage. Total score ranges from 0 to 100, with higher scores representing a better outcome.
Time Frame: Post-Treatment (Week 11)
Measure: Number; unit: percentage who said yes
Arm/Group | Staff Members
Number analyzed (Participants) | 13
percentage who said yes | 100

13. Secondary Outcome: Percent of Staff Who Said They Thought the BRAIN App Would Improve Quality of Life of Persons With Dementia.
Description: Staff were asked if they thought the BRAIN app would improve quality of life of persons with dementia.. The total who said YES was converted into a percentage. Total score ranges from 0 to 100, with higher scores representing a better outcome.
Time Frame: Post-Treatment (Week 11)
Measure: Number; unit: percentage who said yes
Arm/Group | Staff Members
Number analyzed (Participants) | 13
percentage who said yes | 100

ADVERSE EVENTS:
Time Frame: 5 months
Description: Long-term care communities were asked to let the Principal Investigator (PI) know (via email, phone, or in person) about adverse events if/when they occur. In addition, each long-term care community was contacted via email at the end of each month by the PI. In that email, the PI asked the long-term care community whether any adverse events occurred that had not yet been reported. There was no adverse event reporting for staff and family members, as they were not the target of the intervention.
Groups:
- Persons With Dementia: Participants in the Treatment group were invited to participate in one-on-one activity sessions using the Phase 1 version of the BRAIN app twice per week for five weeks.
- Staff Members: Staff members participated by providing feedback on the app and training. In addition, staff took pre- and post-quizzes for the training. NOTE: Staff members were not at risk during the study, because they were not the target of the intervention itself. Instead, they merely provided feedback about the app and took pre and post tests.
- Family Members: Family members exclusively participated by providing information about their loved one's (i.e., person with dementia's) background, interests and preferences. NOTE: Family members were not at risk during the study, because they were not the target of the intervention itself. Instead, they merely provided background information about their loved one.
Arm/Group | Persons With Dementia | Staff Members | Family Members
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/22 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05515679/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05515679/SAP_001.pdf